CLINICAL TRIAL: NCT06013826
Title: University of Health Sciences, Hamidiye Faculty of Nursing
Brief Title: The Effect of Telenursing on the Pain and Fear of Insulin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Associate Proffessor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/0650
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Nurse's Role
Keywords: telenursing, diabetes, pain, fear
MeSH Terms: conditions — Diabetes Mellitus; Pain | interventions — Telenursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients who were randomly assigned to the intervention group were informed about the method of the study. The patient was informed that he would be called before blood glucose measurement and insulin injection for three days to monitor his fear of self-injection and testing. Insulin injection application training was repeated on the first day. Telephone calls made within the scope of tele-health service were recorded in the Telephone Interview Form. During the phone interviews, the questions that the patients wanted to ask were answered. He was asked to fill in the Insulin Injection Evaluation Form according to his experience during the three-day home treatment process. At the end of the three-day meeting, the tele-health service was terminated. D-FISQ was repeated to the patients when they came to the hospital for control.
  Interventions: Other: Telenursing
- Control (No Intervention): Patients who were randomly assigned to the control group were informed about the method of the study. Telehealth service in the control group was not applied. He was asked to fill in the Insulin Injection Evaluation Form according to his experience during the three-day home treatment process. D-FISQ was repeated to the patients when they came to the hospital for control.

INTERVENTIONS:
Other: Telenursing — Patients who were randomly assigned to the intervention group were informed about the method of the study. The patient was informed that he would be called before blood glucose measurement and insulin injection for three days to monitor his fear of self-injection and testing. Insulin injection application training was repeated on the first day. Telephone calls made within the scope of tele-health service were recorded in the Telephone Interview Form. During the phone interviews, the questions that the patients wanted to ask were answered. He was asked to fill in the Insulin Injection Evaluation Form according to his experience during the three-day home treatment process. At the end of the three-day meeting, the tele-health service was terminated.
  Arms: Experimental

SUMMARY:
Aim: The aim of the study is to examine the effects of nursing follow-up with telenursing on the pain and fear factors related to self-injection testing in diabetic individuals who are started on insulin therapy for the first time.

Materials and Methods: The research was implemented in a randomized controlled experimental design. The sample consisted of 70 individuals with diabetes who started insulin therapy for the first time in the diabetes polyclinic of a state university hospital in Istanbul between 17 February and 15 November 2022. Individuals who will start insulin therapy for the first time are directed to the diabetes polyclinic. Insulin Injection Application to all patients in the diabetes polyclinic. In line with the Patient Education Content, the ability to administer insulin, the ability to monitor blood glucose levels, medical nutrition therapy, exercise, etc. applied after the training given on the subjects. Data were collected with the Patient Information Form, Diabetic Self-Injection and Fear of Testing Questionnaire Form (D-SFIQ), Insulin Injection Evaluation Form. Patients assigned to the intervention group were given telehealth service for three days for fear of self-injection and testing.

DETAILED DESCRIPTION:
The sample of the study consisted of 70 patients who met the inclusion criteria and agreed to participate. Insulin therapy was evaluated according to the inclusion criteria and those who agreed to participate in the study. 19 doctors and 2 nurses work in the diabetes polyclinic. Individuals who will start insulin therapy for the first time after a doctor's examination are referred to the diabetes polyclinic. The history of the patients who come to the diabetes polyclinic is taken by the diabetes nurse and their physical examination is performed. In the diabetes polyclinic, all patients are taught by the diabetes education nurse, the ability to administer insulin, the ability to monitor blood glucose levels, medical nutrition therapy, exercise, etc. subjects are taught. After the training, the patients are called for control seven days later. However, a nursing follow-up is not applied during this process until it comes to control again. In our study, all patients were given training on insulin administration and testing by subcutaneous route using the Insulin Injection Application Patient Education Content, accompanied by a diabetes polyclinic nurse. In line with the content of the training, it was applied in the form of explaining to all patients with the subcutaneous injection application model, answering the questions of the patients or their relatives with the question-answer method, monitoring the patient while practicing on the model by the researcher, and repeating the training in line with the needs. After the training, all patients who accepted to participate in the study were recorded with the Patient Information Form, as well as their individual characteristics and information about the disease and treatment characteristics. D-FISQ was applied by the face-to-face interview method. The application of the study was continued according to the groups to which they were assigned by randomization (Figure 3.1).

Experimental group intervention Patients who were randomly assigned to the intervention group were informed about the method of the study. The patient was informed that participant would be called before blood glucose measurement and insulin injection for three days to monitor his fear of self-injection and testing. Insulin injection application training was repeated on the first day. Telephone calls made within the scope of tele-health service were recorded in the Telephone Interview Form. During the phone interviews, the questions that the patients wanted to ask were answered. The topics that the patients most frequently asked for support are listed in Table 1. The participant was asked to fill in the Insulin Injection Evaluation Form according to his experience during the three-day home treatment process. At the end of the three-day meeting, the tele-health service was terminated. D-FISQ was repeated to the patients when they came to the hospital for control.

Control group intervention Patients who were randomly assigned to the control group were informed about the method of the study. Telehealth service in the control group was not applied. The participant was asked to fill in the Insulin Injection Evaluation Form according to his experience during the three-day home treatment process. D-FISQ was repeated to the patients when they came to the hospital for control.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Absence of physical, mental inadequacy and communication difficulties,
* Having a diagnosis of type II diabetes,
* Initiation of insulin therapy for the first time,
* Measuring blood sugar at least once a day,
* Self-administration of insulin injection,
* Ability to communicate by phone,
* Not having administered a self-injection of insulin before.

Exclusion Criteria:

* Having physical, mental inadequacy and communication difficulties,
* Having a history of allergy,
* Being pregnant,
* Not starting insulin therapy for the first time,
* Not measuring blood sugar at least once a day,
* Not self-administering insulin injection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Injection Pain | Through study completion, an average of 1 months
  In order to identify the pain that occurs during insulin injection in patients, Insulin injection evaluation form was used. The form created by the researcher was used to determine the difficulties that patients face while administering insulin injections. The form consists of a total of 3 sections and 18 questions regarding the presence of pain, finger puncture pain intensity, drug administration pain intensity, injection administration difficulty, insulin dose skipping.
  In order to evaluate the items in the form in terms of relevance and scope, it was submitted to the opinion of 4 experts working in the unit and working as educators in undergraduate and graduate programs. After the expert opinion, the items were reviewed and the form was finalized in line with the suggestions.
Fear | Through study completion, an average of 1 months
  The Diabetes Fear of Self Injecting and Self-testing Questionnaire-D-FISQ was used to define the fear of self-injection and testing in diabetics. The validity and reliability of the D-FISQ developed by Snoek et al. (1997) for the Turkish population was performed by Çelik and Pınar (2016). D-FISQ, which includes 15 statements, consists of two sub-dimensions: fear of self-injecting (fear of self-injecting-FSI, 6 statements) and fear of self-testing (fear of self-testing-FST, 9 statements).

CONTACTS AND LOCATIONS:
Overall Officials: Demet İnangil, Study Chair — Saglik Bilimleri Universitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Demet İnangil, Istanbul
  - Saglik Bilimleri University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Souza-Junior VD, Mendes IA, Mazzo A, Godoy S. Application of telenursing in nursing practice: an integrative literature review. Appl Nurs Res. 2016 Feb;29:254-60. doi: 10.1016/j.apnr.2015.05.005. Epub 2015 May 20. PMID 26856523
- [Background] Peng X, Su Y, Hu Z, Sun X, Li X, Dolansky MA, Qu M, Hu X. Home-based telehealth exercise training program in Chinese patients with heart failure: A randomized controlled trial. Medicine (Baltimore). 2018 Aug;97(35):e12069. doi: 10.1097/MD.0000000000012069. PMID 30170422